CLINICAL TRIAL: NCT03823209
Title: Increasing PrEP Use in High-Risk Social Networks of African-American MSM in Underserved Low-Risk Cities
Acronym: SNAP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Jeffrey Kelly, Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PRO00029359
Record Dates: First submitted 2019-01-24; First posted 2019-01-30 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Human Immunodeficiency Virus
Keywords: Pre-exposure prophylaxis (PrEP)
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social Network Approach (Experimental): Participants will receive brief HIV counseling at baseline visit.
  Leaders of social networks will be determined using data from participants. These leaders will then be invited to attend a 5-session small-group training that will teach them how to communicate the benefits of PrEP to their social network members.
  All social network members will be asked about intervention exposure at 6- and 15-month followups.
  Interventions: Behavioral: Social Network; Behavioral: Brief HIV Prevention Counseling
- Comparison (Active Comparator): Participants will receive brief HIV counseling at baseline visit.
  Interventions: Behavioral: Brief HIV Prevention Counseling

INTERVENTIONS:
Behavioral: Social Network — Leaders of social networks will be statistically determined. Over 5 small-group training sessions, these leaders will be trained to communicate to their social network members accurate information about PrEP and its availability; correct PrEP misconceptions and negative stereotypes; endorse PrEP use and its benefits; and strengthen friends' attitudes, intentions, perceived peer norms, and self-efficacy regarding PrEP as a personal HIV protective strategy.
  Arms: Social Network Approach
Behavioral: Brief HIV Prevention Counseling — Participants will receive brief (15-minute) counseling on how to prevent HIV infection.

SUMMARY:
This study evaluates the use of a social-network approach to encourage African-American men who have sex with men (AAMSM) to adopt pre-exposure prophylaxis (PrEP) to prevent HIV infection. Thirty-six networks of AAMSM will be recruited in Milwaukee, WI, and Cleveland, OH. Half of these networks will have their leaders trained to endorse PrEP to their social network members, and the other half will be given brief HIV prevention counseling.

DETAILED DESCRIPTION:
Pre-exposure prophylaxis (PrEP) regimens greatly reduce the likelihood that high-risk uninfected men who have sex with men (MSM) will contract HIV infection. Although this protective benefit has been unequivocally established in clinical trials, the number of high-risk men on PrEP remains far below the threshold needed to substantially reduce HIV incidence. This is especially true outside of the country's largest cities. Novel approaches are needed to increase PrEP use among high-risk racial minority MSM in these neglected cities.

This study will recruit 36 sociocentric social networks of high-risk young racial minority MSM, 18 networks per city (total n=36 networks x 14 anticipated recruited members per network = 504 participants). Participants will complete measures assessing baseline PrEP use; knowledge, attitudes, perceived norms, intentions, and stage of readiness for PrEP; sexual risk practices and substance use; and prior or current ART use. Participants will also complete measures used to identify each network's leaders.

Networks will be randomized in equal numbers in each city to comparison or intervention conditions. All study participants will receive individual baseline counseling about risk reduction and PrEP, with referral offered to clinics prescribing PrEP. Members of the 18 experimental condition networks will also receive the social network PrEP intervention being tested in the study. In it, cadres of leaders in each network-selected based on their leadership position within the network and their own openness to PrEP-will attend a 5-session intervention that trains, engages, and supports network leaders in communicating to friends accurate information about PrEP and its availability; corrects PrEP misconceptions and negative stereotypes; endorses PrEP use and its benefits; and strengthens friends' attitudes, intentions, perceived peer norms, and self-efficacy regarding PrEP as a personal HIV protective strategy. Two additional booster sessions spaced monthly will support maintenance of leaders' efforts in talking with friends in their network about the benefits of PrEP, as well as where and how to access it.

At 6- and 15-month followup points, all study participants will complete the same behavioral measures that were administered at baseline, as well as measures of intervention exposure.

ELIGIBILITY:
Inclusion Criteria:

INDIVIDUALS:

1. Age 16 or older
2. For the seed only, self-report of HIV-negative serostatus or unknown serostatus
3. Except for the seed, being named as a friend by an already-enrolled participant
4. Male at birth
5. Sex with at least one male partner in the past 12 months

NETWORKS

1. More than 49% of the seed's eligible friends agree to participate
2. More than 49% of all network members self-report they are HIV-negative at baseline

Exclusion Criteria:

INDIVIDUALS:

1. Age 15 or younger
2. For the seed only, self-report of HIV-positive serostatus
3. Except for the seed, not being named as a friend by an already-enrolled participant
4. Not male at birth
5. No report of sex with at least one male partner in the past 12 months

NETWORKS

1. Less than 50% of the seed's eligible friends agree to participate
2. Less than 50% of all network members self-report they are HIV-negative at baseline

Min Age: 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2019-01-24 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Self-report of pre-exposure prophylaxis (PrEP) use | 6 and 15 months
  Change in self-reported PrEP use

SECONDARY OUTCOMES:
Pre-Exposure Prophylaxis (PrEP) Knowledge | 6 and 15 months
  PrEP Knowledge: 13 items in scale, items are added to determine score, with higher scores indicating greater knowledge
  Scale taken from Walsh, J.L. (2018). Applying the Information-Motivation-Behavioral Skills Model to Understand PrEP Intentions and Use Among Men Who Have Sex with Men. AIDS and Behavior.
Pre-Exposure Prophylaxis Attitudes | 6 and 15 months
  PrEP Attitudes: 5 items in scale, items are averaged to determine score, with higher scores indicating more positive attitudes
  Scale taken from Walsh, J.L. (2018). Applying the Information-Motivation-Behavioral Skills Model to Understand PrEP Intentions and Use Among Men Who Have Sex with Men. AIDS and Behavior.
Pre-Exposure Prophylaxis Norm Perceptions | 6 and 15 months
  PrEP Norm Perceptions: 6 items in scale, items are averaged to determine score, with higher scores indicating more favorable norms
  Scale taken from Walsh, J.L. (2018). Applying the Information-Motivation-Behavioral Skills Model to Understand PrEP Intentions and Use Among Men Who Have Sex with Men. AIDS and Behavior.
Pre-Exposure Prophylaxis Intentions | 6 and 15 months
  PrEP Intentions: 3 items in scale, items are averaged to determine score, with higher scores indicating greater intentions to use PrEP
  Scale taken from Walsh, J.L. (2018). Applying the Information-Motivation-Behavioral Skills Model to Understand PrEP Intentions and Use Among Men Who Have Sex with Men. AIDS and Behavior.
Pre-Exposure Prophylaxis Self-Efficacy | 6 and 15 months
  PrEP Self-Efficacy: 8 items in scale, items are averaged to determine score, with higher scores indicating greater self-efficacy for PrEP use.
  Scale taken from Walsh, J.L. (2018). Applying the Information-Motivation-Behavioral Skills Model to Understand PrEP Intentions and Use Among Men Who Have Sex with Men. AIDS and Behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A. Kelly, PhD, Principal Investigator — Medical College of Wisconsin; Yuri A. Amirkhanian, PhD, Principal Investigator — Medical College of Wisconsin
Locations (2):
- United States (2):
  - AIDS TaskForce of Greater Cleveland, Cleveland, Ohio
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kelly JA. Ten Things We Need to Do to Achieve the Goals of the End the HIV Epidemic Plan for America. J Acquir Immune Defic Syndr. 2019 Dec 1;82 Suppl 2(2):S94-S98. doi: 10.1097/QAI.0000000000002166. PMID 31658194
- [Result] Quinn KG, Christenson E, Spector A, Amirkhanian Y, Kelly JA. The Influence of Peers on PrEP Perceptions and Use Among Young Black Gay, Bisexual, and Other Men Who Have Sex with Men: A Qualitative Examination. Arch Sex Behav. 2020 Aug;49(6):2129-2143. doi: 10.1007/s10508-019-01593-x. Epub 2020 Feb 3. PMID 32016815
- [Result] Kelly JA, Amirkhanian YA, Walsh JL, Brown KD, Quinn KG, Petroll AE, Pearson BM, Rosado AN, Ertl T. Social network intervention to increase pre-exposure prophylaxis (PrEP) awareness, interest, and use among African American men who have sex with men. AIDS Care. 2020 May;32(sup2):40-46. doi: 10.1080/09540121.2020.1739207. Epub 2020 Mar 13. PMID 32167374

DOCUMENTS (1):
  • Informed Consent Form (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT03823209/ICF_000.pdf